CLINICAL TRIAL: NCT05416346
Title: The Feasibility and Effectiveness of Digital Cognitive Behavioral Therapy for Insomnia in China: A Pilot Randomized Controlled Trial
Brief Title: Digital Cognitive Behavioral Therapy for Insomnia in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: dCBT-i-Chinese
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Primary Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dCBT-i (Experimental): The dCBT-i group received the whole intervention
  Interventions: Behavioral: Digital Cognitive Behavioral Therapy
- Sleep Hygiene Education (SHE) (Active Comparator): The SHE group received sleep hygiene education delivered in text form, and the same intervention as the dCBT-i group did after four weeks.
  Interventions: Behavioral: Digital Cognitive Behavioral Therapy; Behavioral: Sleep Hygiene Education (SHE)

INTERVENTIONS:
Behavioral: Digital Cognitive Behavioral Therapy — Cognitive behavioral therapy for insomnia (CBT-i) has been showed to be effective in reducing insomnia symptoms and insomnia-related symptoms, including sleepiness, dysfunctional beliefs and attitudes about sleep, anxiety and depressive symptoms
Behavioral: Sleep Hygiene Education (SHE) — The SHE group received sleep hygiene education delivered in text form, and the same intervention as the dCBT-i group did after four weeks.
  Arms: Sleep Hygiene Education (SHE)

SUMMARY:
Digital cognitive behavioral therapy for insomnia (dCBT-i) is found to be effective but is rarely used in China. Hence, the investigators developed an automated Chinese dCBT-i program and examined its feasibility, acceptability, and preliminary effectiveness in individuals with insomnia symptoms.

ELIGIBILITY:
Inclusion Criteria:

* were aged 18 or older;
* had a positive screening result for chronic insomnia, i.e., a score of 16 or lower on the Sleep Condition Indicator (SCI);
* had stable access to the internet via a smartphone.

Exclusion Criteria:

* additional sleeping conditions except for insomnia (such as restless legs syndrome and sleep apnea);
* psychosis or mania;
* serious physical health concerns necessitating surgery or with prognosis <6 months;
* undergoing medical or psychological treatment for insomnia with a health professional;
* habitual night shift, evening, or rotating shift-workers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2021-06-12 (Actual)

PRIMARY OUTCOMES:
sleep diary | week 4
  recording one's sleep efficiency, total sleep time, sleep onset latency, wakefulness after sleep onset, and subjective sleep quality
Sleep Condition Indicator-8 | week 4
  Sleep Condition Indicator-8 is an 8-item scale validated against Diagnostic and Statistical Manual-5 criteria, concerning sleep quality and daytime personal functioning. It scores between 0 to 32, with higher scores meaning better sleep.

SECONDARY OUTCOMES:
the Insomnia Severity Index 7-item version | week 4
  It scores between 0 to 28, with higher scores meaning more severe insomnia.
the Dysfunctional Beliefs and Attitudes about Sleep Scale 16-item version | week 4
  It scores between 16 to 80, with higher scores meaning more dysfunctional beliefs.
the Epworth Sleepiness Scale | week 4
  It scores between 0 to 24, with higher scores meaning greater sleepiness.
the Patient Health Questionnaire 9-item version | week 4
  It scores between 0 to 27, with higher scores meaning higher depressive symptoms.
the Generalized Anxiety Disorder 7-item version | week 4
  It scores between 0 to 21, with higher scores meaning higher anxious symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided